CLINICAL TRIAL: NCT06573385
Title: Evaluation of Validity and Reliability of the Turkish Version of the Diabetes Education Questionnaire (DATE-Q) in Patients with Diabetes
Brief Title: Reliability and Validity of Turkish Version of the Diabetes Education Questionnaire (DATE-Q)
Status: Completed | Type: Observational
Sponsor: Biruni University (Other)
Collaborators: Istanbul University (Other); Istanbul Galata University (Other)
Responsible Party: Principal Investigator, Buket AKINCI, Assoc. Prof., Biruni University
Other Study IDs: 2024/1193
Record Dates: First submitted 2024-08-24; First posted 2024-08-27 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Questionnaire — Questionnaire application

SUMMARY:
The Diabetes Education Questionnaire (DATE-Q) is a questionnaire that includes comprehensive care components of diabetes management and specifically questions the effect of exercise on blood glucose levels and the knowledge of the correct exercise intensity in patients with diabetes. It can be easily and rapidly applied. The aim of this study is to evaluate the translation into Turkish, validity and reliability of the DATE-Q, which questions the knowledge of diabetic patients about their disease.

ELIGIBILITY:
Inclusion Criteria:

. Age of 18 or above

* Those whose native language is Turkish
* Volunteer to participate in the study

Exclusion Criteria:

* Individuals who cannot cooperate (those who score below 24 points according to the Standardized Mini Mental Test)
* Those who have problems understanding and speaking Turkish
* Any visual or cognitive disorder that would prevent the participant from answering the survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients who are diagnosed with Diabetes
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Diabetes Education Questionnaire (DATE-Q) | Day 1
  The Diabetes Education Questionnaire (DATE-Q) is a questionnaire that includes comprehensive care components of diabetes management and specifically questions the effect of exercise on blood glucose levels and the knowledge of the correct exercise intensity in patients with diabetes. The questionnaire was designed to be a true/false/I don't know questionnaire, with 20 items (four in each domain). With each correct answer as 1 point, the maximum score possible is 20 overall, 4 by domain.

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni Üniversitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No